CLINICAL TRIAL: NCT05238012
Title: A 24-week, Multi-center, Randomized, Open-Label Clinical Trial to Compare the Impact of Xuezhikang and Atorvastatin on Glucose Metabolism in Dyslipidemia Patients With Prediabetes (XTREME Study)
Brief Title: Compare the Impact of Xuezhikang and Atorvastatin on Glucose Metabolism in Dyslipidemia Patients With Prediabetes
Acronym: XTREME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heart Health Research Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-21-21279
Record Dates: First submitted 2022-01-14; First posted 2022-02-14 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Metabolism Disorder, Lipid; Metabolism Disorder, Glucose
Keywords: Dyslipidemia; Prediabetes
MeSH Terms: conditions — Lipid Metabolism Disorders; Glucose Metabolism Disorders; Dyslipidemias; Prediabetic State | interventions — xuezhikang; Atorvastatin

STUDY DESIGN:
Intervention Model Description: Experimental group: Xuezhikang Capsule, 1200mg / day, twice a day, 2 capsules each time, after meals in the morning and evening.
  Control group: Atorvastatin Calcium Tablets, 20mg/day, once a day, one tablet each time, before bedtime; Continuous treatment for 24 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xuezhikang Capsule (Experimental): Experimental drug: Xuezhikang Capsule, specification: 300mg / capsule.
  Interventions: Drug: Xuezhikang Capsule
- Atorvastatin Calcium Tablets (Active Comparator): Control drug: Atorvastatin Calcium Tablets, specification: 20mg / tablet.
  Interventions: Drug: Atorvastatin Calcium Tablets

INTERVENTIONS:
Drug: Xuezhikang Capsule — Xuezhikang Capsule, 1200mg / day, twice a day, 2 capsules each time, after meals in the morning and evening.
  Arms: Xuezhikang Capsule
Drug: Atorvastatin Calcium Tablets — Atorvastatin Calcium Tablets, 20mg/day, once a day, one tablet each time, before bedtime;
  Arms: Atorvastatin Calcium Tablets

SUMMARY:
This study is a prospective, randomized, open-label, multi-center trial. The primary objective of the study is to assess whether XZK 1200mg/d, compared to atorvastatin 20mg/d, has a favorable impact on HbA1c levels at 24 weeks of treatment in dyslipidemia patients with prediabetes

DETAILED DESCRIPTION:
Up to now, there is no published RCTs to compare the impact of XZK and statins on glucose metabolism in Prediabetes with dyslipidemia. However, systematic reviews of several large observational studies have recently found statin treatment is associated with a modest increase in HbA1c in patients with T2DM. In these patients, the mean difference of HbA1c increased by 0.17% (95% CI 0.07, 0.27) compared with the blanking control group[7]. For instance, Atorvastatin 20mg is widely used medium intensity statin in clinical practice, but a cohort study based on a database of Korea populations reported that the use of low dose Atorvastatin 10-20mg tended to be a risk factor for onset diabetes (NODM) in Asians[8]. Meanwhile, a small RCT reported that HbA1c level was increased from 6.1% to 6.5% after Atorvastatin 20mg/d treatment for 2 months[9]. The long-term administration of statins might increase the risk of NODM approximately 10%-12%[10]. In short, a diabetogenic role of statins has been demonstrated both from randomized trials and meta-analyses, and risk factors include high dose, prolonged exposure, old age, prediabetic state and metabolic syndrome[11, 12]. In consideration of prediabetes, including IFG, IGT, or A1C 5.7-6.4%, will be further increased the risk of development diabetes mellitus, and the prevalence was 35.7% in China, we choose the patients in Prediabetes with dyslipidemia in our study[4].

XZK, a partially purified red yeast rice (RYR) under controlled pharmaceutical manufacturing conditions, contains a family of naturally occurring statins (monacolins)-most prominently monacolin K, which is identical to the lipid- lowering therapy lovastatin (Mevacor)[13]. In a meta-analysis, after compared the XZK treatment group showed significant lowering LDL-C effect compared with basic therapy groups. [14] Xuezhikang in the China Coronary Secondary Prevention Study trial(CCSPS) has shown that XZK significantly reduced the levels of TC, TG and LDL-C and increased that of HDL-C in patients with hyperlipidemia after 1200mg/d treatment for 8 weeks, among which TC decreased by 23.0%[15]. Furthermore, a retrospective cohort study that used Taiwan's National Health Insurance data on 34,504 persons with a RYR prescription in 2010-2014, found that a lower risk of incident diabetes when compared to lovastatin cohort (HR:0.46, 95% CI 0.43-0.50)[16]. Why XZK can lower the risk of incident diabetes compared to other statins? A variety of mechanisms have been elucidated. As main components in XZK, n-3 polyunsaturated fatty acid(PUFAs) can regulate the activity of key transcription factors to regulate gene expression in lipid metabolism and improve insulin sensitivity of type 2 diabetes mellitus to prevent diabetic complications. Six weeks of supplementation with n-3 PUFAs reduced the postprandial decrease in macrovascular function and meanwhile improved postprandial microvascular function[17]. Moreover, it was reported that magnesium deficiency can lead to the reduction of insulin sensitivity and affect the stability of glucose metabolism. Thus, increasing the intake of magnesium plays an important role in the prevention of noninsulin- dependent diabetes mellitus and its complications. Moreover, selenium reduces the production of oxygen free radicals in the body by glutathione peroxidase to prevent further oxidative damage in the body and the insulin A, B between the two peptide chains for ensuring the complete molecule structure and function of insulin to play a role in lowering blood glucose. In addition, selenium also has inhibitory effects on complications of diabetes such as osteoporosis and retinopathy.

In addition, XZK has been proved to contain multiple active ingredients which leads to unique MOA and multiple benefits[13]. It is composed of 13 kinds of natural statins, unsaturated fatty acids, ergosterol, amino acids, flavonoids, alkaloid, trace elements, and other substances, and thus could be regarded as a natural lipid lowering polypill[14]. All the above-mentioned components might be involved in the mechanism of XZK to multiple benefits such as antiatherosclerosis, liver protection, anticancer, neural regulation and protection, and kidney protection effects[13]. Previous animal and cell experiments have shown that XZK can also activate the PPARα pathway and up-regulate apolipoprotein A5 (apolipoprotein A5 is the key regulator of TG metabolism) to achieve higher TG reduction when it reduces LDL-C by the same extent as simvastatin[18]. It is speculated that non-statin elements within XZK may play a synergistic role in regulating blood lipids and inhibiting the synthesis of triglycerides. The China Coronary Secondary Prevention Study (CCSPS) and other clinical studies confirmed that XZK capsules reduce lipid and significantly reduce the overall mortality of patients with coronary heart disease, the incidence of cardiovascular events. According to Chinese guidelines for the management of dyslipidemia in adults of 2016 revision, XZK amongst other statins are recommended for the first-line treatment of cholesterol controlling. Meanwhile, XZK 1200mg/d and Atorvastatin 20mg/d are medium intensity statins recommended in guideline[3]. therefore, we choose Atorvastatin 20mg/d as control drug in our research.

Physicians faced with a dyslipidemia patient with prediabetes often use statins therapy due to perceived efficacy. However, XZK is a promising option in this patient group due to their significantly lower risk of dys-glycaemia without compromising efficacy for lowering lipids in hyperlipidemia. Establishing comparable recurrent NODM rates in individuals with previous Prediabetes state would result in superior DM prevention for these patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent provided
* 2. Age ≥40 years
* 3 Diagnosed Prediabetes, meeting one of the following conditions: ü Impaired fasting glucose (IFG): 5.6 mmol/L ≤ FPG <7.0 mmol/L ; ü HbA1c 5.7-6.4% (39-47 mmol/mol)
* 4. Dyslipidemia meets one of the following conditions: ü Fasting LDL-C ≥3.4mmol/L and<4.9mmol/L，and TG≤5.6 mmol/L ü Fasting non-HDL-C ≥4.1mmol/L and < 5.7 mmol/L , and TG≤5.6 mmol/L
* 5. Completed one-week Patient diary, recorded at least 5 days in a week.

Exclusion Criteria:

* 1. Patient with proven or documented atherosclerotic cardiovascular disease (ASCVD), including acute coronary syndrome (ACS), history of myocardial infarction (MI), stable or unstable angina pectoris, coronary or other revascularization, ischemic stroke, transient ischemic attack and peripheral vascular disease (PAD), etc.
* 2.Diagnosed diabetes According to 2021 the American Diabetes Association (ADA) "Standards of Medical Care in Diabetes" FPG≥126mg/dL(7.0mmol/L). A know 2-hPG≥200mg/dL(11.1mmol/L)duringOGTT. A1C≥6.5%(48mmol/mol). In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥200 mg/dL (11.1 mmol/L).
* 3. Patientswithanylipidloweringdrugsintheprevious3months,includingbut not limited to statins, bile acid sequestrants, cholesterol absorption inhibitors, PCSK9 inhibitors, nicotinic acid, fibric acid derivatives, fibrates, other traditional Chinese medicine and n-3 fatty acids.
* 4.Patientswithanyantidiabeticdrugs.
* 5.ContraindicationstoXZKorAtorvastatin: Allergic to XZK or Atorvastatin. Pregnancy or breastfeeding
* 6.Uncontrolled hypertension (systolic blood pressure ≥180 mm Hg and/ or diastolic blood pressure ≥110 mm Hg) at screening.
* 7.Active liver disease or hepatic dysfunction, including continuously elevated liver transaminase due to unknown causes. Abnormal liver function test at baseline (ALT or AST >3×ULN).
* 8. Knownrenaldysfunctionorelevatedserumcreatininelevelsatbaseline(with an eGFR≤60 mL/min/1.73 m2).
* 9.Otherendocrinediseasesthatmightinfluencethelevelsoflipidorlipoprotein, such as hypothyroidism.
* 10.Patient has participated in clinical trials of other drugs in the past three months.
* 11.Previous statin treatment causes creatine kinase (CK) increased 10 times, or myalgia myopathy (muscle pain or muscle weakness, accompanied by Creatine phosphokinase (CK) exceeds 10 times the ULN)
* 12.Estimated life expectancy < 6 months at the time of enrollment
* 13.Abuse of alcohol, or history of alcohol abuse.
* 14.Close affiliation with the investigators, e.g., a close relative for the investigator, dependent person (e.g., employee or student of the investigators)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
HbA1c levels | 24 weeks
  To determine whether XZK 1200mg/d, compared to atorvastatin 20mg/d, has a favorable impact on HbA1c levels from baseline to 24 weeks in dyslipidemia patients with prediabetes.

SECONDARY OUTCOMES:
Fasting blood glucose(FBG), | 24 weeks
  The change value of FBG from baseline to 24 Weeks or before antidiabetic therapy initiation within 24 weeks.
Post prandial glucose(PPG) 2h | 24 weeks
  The change value of PPG 2h from baseline to 24 Weeks or before antidiabetic therapy initiation within 24 weeks.
HOMA-IR | 24 weeks
  The change value of HOMA-IR from baseline to 24 Weeks or before antidiabetic therapy initiation within 24 weeks.
LDL-C levels | 24 weeks
  The percentage change of LDL-C levels from baseline to 24 Weeks or before antidiabetic therapy initiation within 24 weeks.
non HDL-C levels | 24 weeks
  The percentage change of non HDL-C levels from baseline to 24 Weeks or before antidiabetic therapy initiation within 24 weeks.
HbA1c levels | 12 Weeks
  The change value of HbA1c levels from baseline to 12 Weeks or before antidiabetic therapy initiation within 12 weeks.
Fasting blood glucose(FBG) | 12 weeks
  The change value of FBG from baseline to 12 Weeks or before antidiabetic therapy initiation within 12 weeks.
Post prandial glucose(PPG) 2h | 12 weeks
  The change value of PPG 2h from baseline to 12 Weeks or before antidiabetic therapy initiation within 12 weeks.
HOMA-IR | 12 weeks
  The change value of HOMA-IR from baseline to 12 Weeks or before antidiabetic therapy initiation within 12 weeks.
LDL-C levels | 12 weeks
  The percentage change of LDL-C levels from baseline to 12 weeks or before antidiabetic therapy initiation within 12 weeks.
non HDL-C levels | 12 weeks
  The percentage change of non HDL-C levels from baseline to 24 Weeks or before antidiabetic therapy initiation within 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

DOCUMENTS (1):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT05238012/Prot_000.pdf